CLINICAL TRIAL: NCT03002909
Title: Effect of Continuous Pre-peritoneal Wound Infiltration Versus Epidural Analgesia on Inflammatory Response and Pain Following Radical Cytsectomy
Brief Title: Continuous Pre-peritoneal Wound Infiltration Versus Epidural Analgesia in Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif,MD, lecturer of anesthesia ,icu and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 369
Record Dates: First submitted 2016-12-19; First posted 2016-12-26 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2017-12

CONDITIONS: Abdominal Neoplasms
MeSH Terms: conditions — Abdominal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- epidural group (Active Comparator): an epidural catheter will be inserted under sterile conditions through the T9- 12 interspace using the 'loss-of-resistance' technique. The catheter will be advanced 4 cm cephalad. .
  Interventions: Device: epidural catheter
- preperitoneal group (Active Comparator): preperitoneal catheters will be placed in the subfascial (ie, pre-peritoneal) space under direct vision.
  Interventions: Device: preperitoneal catheter

INTERVENTIONS:
Device: epidural catheter
  Other Names: PEA block
  Arms: epidural group
Device: preperitoneal catheter
  Other Names: preperitoneal infusion
  Arms: preperitoneal group

SUMMARY:
the investigators aim is to investigate the effect of continuous preperitoneal bupivacaine wound infiltration versus epidural analgesia on the inflammatory cytokines response following radical cytectomy

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* aged 18-60 yr
* undergo open abdominal cancer surgery

Exclusion Criteria:

* general contraindications for epidural analgesia,
* recent history (8 weeks) of, chemotherapy or radiation,
* chronic opioid use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01; Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
changes in the level of inflammatory cytokines in pg /ml | 24 hours
  Blood samples taken all over the 24-hr. period were collected in plasma tubes containing ethyl-enediamine-tetra-acectic (EDTA), centrifuged and stored at 20○c for assessment of Plasma concentrations plasma IL 1, IL 6, IL10 and TNF to assess inflammatory cytokines

SECONDARY OUTCOMES:
Visual Analog Scale at rest and on coughing | 24 hours
  pain intensity was assessed using a 10-cm VAS (0 = no pain and 10 = worst imaginable pain)
opioid side-effects | 24 hours
  observation of side effects and record incidence as nausea, vomiting and itching
patient satisfaction | 24 hours
  scale ranging 1-4 :unsatisfactory, regular, satisfactory and excellent)

CONTACTS AND LOCATIONS:
Overall Officials: fatma el sherif, M.D, Principal Investigator — south Egypt cancer institute - assuit university; Ahmad M Abd El-Rahman, M.D, Study Director — Lecturer of anesthesia, icu, and pain management
Locations (1):
- South Egypt Cancer instIitute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Othman AH, Ahmed DG, Abd El-Rahman AM, El Sherif FA, Mansour S, Aboeleuon E. Effect of Preperitoneal Versus Epidural Analgesia on Postoperative Inflammatory Response and Pain Following Radical Cystectomy: A Prospective, Randomized Trial. Clin J Pain. 2019 Apr;35(4):328-334. doi: 10.1097/AJP.0000000000000679. PMID 30829734